CLINICAL TRIAL: NCT04532138
Title: A Comparison Between C-MAC Video Laryngoscope an VS-CMAC Rigid Fiberoptic Stylet for Awake Endoscopic Intubation in Severe Predicted Difficult Airways: a Randomized Controlled Trial
Brief Title: C-MAC Video Laryngoscope and VS-CMAC Fiberoptic Stylet for Awake Endoscopic Intubation in Predicted Difficult Airways
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Director of the Clinic of Anaesthesia and Intensive Care, Principal Investigator, Clinical Professor, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D-BLADE - VS
Record Dates: First submitted 2020-07-21; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Difficult Airway Intubation
Keywords: difficult airway; difficult intubation; awake endoscopic intubation; rigid fiberoptic stylet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C-MAC Video laryngoscope awake intubation (Active Comparator): In this group, patients with severe predicted difficult airways scheduled for elective surgery receive awake endoscopic intubation using Videolaryngoscope (C-MAC) with Hyperangulated blade (D-blade) Spontaneous breathing will be preserved in both groups of patients enrolled and the same protocol of sedation plus upper airways topical anesthesia will be applied.
  Interventions: Device: C-MAC Video laryngoscope awake intubation
- VS-CMAC Rigid Fiberoptic Stylet awake intubation (Experimental): In this group, patients with severe predicted difficult airways scheduled for elective surgery receive awake endoscopic intubation using VS-CMAC Rigid Fiberoptic Stylet.
  Spontaneous breathing will be preserved in both groups of patients enrolled and the same protocol of sedation plus upper airways topical anesthesia will be applied.
  Interventions: Device: VS-CMAC Rigid Fiberoptic Stylet

INTERVENTIONS:
Device: VS-CMAC Rigid Fiberoptic Stylet — patients with severe predicted difficult airways scheduled for elective surgery randomized to this groups will receive awake endoscopic intubation using VS-CMAC Rigid Fiberoptic Stylet.
  Arms: VS-CMAC Rigid Fiberoptic Stylet awake intubation
Device: C-MAC Video laryngoscope awake intubation — patients with severe predicted difficult airways scheduled for elective surgery randomized to this groups will receive awake endoscopic intubation using C-MAC Video Laryngoscope intubation.
  Other Names: videolaryngoscope with hyperangulated blade
  Arms: C-MAC Video laryngoscope awake intubation

SUMMARY:
An Anticipated difficult tracheal intubation is recommended to be managed performing the so called "Awake tracheal endoscopic intubation" (ATI) with the maintenance of patient's spontaneous breathing after an adequate sedation and topical anesthesia of upper airways, providing supplemental oxygen.

Initially only flexible bronchoscope was considered the device of choice (the gold standard) for ATI but in the last decade videolaryngoscopes with hyper-angulated blade have been demonstrated to be an efficacy technique.

Most recently, endoscopic rigid stylets such as Bonfils (Carl Storz™) and Sensacope (Acoutronic™) have been proposed as alternative techniques for ATI in the event of expected difficult tracheal intubation.

However, to date, no comparison studies have been carried out between these two kind of devices, alternative to flexible fiberscope, for ATI.

This is a clinical prospective randomized-controlled trial of non inferiority. The aim of this study is to compare the intubation success rate between two different devices (C-MAC Video Laryngoscope and VS-CMAC fiberoptic stylet) in patients with severe predicted difficult airways scheduled for elective surgery.

The primary endpoint is the comparison of success rate for the tracheal intubation, demonstrating the non inferiority of videostylet efficacy compared to the most consolidated technique based on videolaryngoscope.

DETAILED DESCRIPTION:
This is a clinical prospective randomized-controlled trial of non inferiority, set in the operating theatre of a terziary university hospital in Ancona (Ospedali Riuniti Ancona).

The aim of this study is to compare the intubation success rate, defined as correct positioning of the tracheal tube inside the trachea, between Videostylet (VS-Carl Storz™) and videolaryngoscope with hyperangulated blade (C-MAC - Carl Storz™) in patients with severe predicted difficult airways scheduled for elective surgery.

All patients enrolled in the study, examined in the pre-operative visit, will be asked for informed consent and will undergo the same anesthetic protocol consisting in upper airways topicalization with Lidocaine and in smooth/moderate sedation (targeted on Ramsay sedation scale ≦ 3) by i.v. administration of midazolam 0,03 mg/kg and Fentanyl 100 mcg.

On arrival in the operating room, nasal oxygen (5 L/min) and routine monitoring of vital signs will be applied to all patients.

Heart rate and blood pressure will be recorded at the beginning of the procedure and every 3 minutes until the intubation will be performed, while arterial oxygen saturation is continuously recorded.

Patients enrolled will be randomly divided into 2 groups regarding to the device used for ATI:

1. Videolaryngoscope (C-MAC) with Hyperangulated blade (D-blade)
2. Videostylet (VS) Endotracheal tube will be 6,5-7,0 mm for female and 7,5-8,0 mm for male.

The following parameters will be registered:

* success rate of the procedure defined as correct positioning of the tracheal tube in the trachea confirmed both endoscopically and through the capnographic curve EtCO2
* average time of intubation procedure expressed in sec.
* operator's assessment of the subjective difficulty / handling of the device by means of a special analogue numerical scale
* assessment of the patient's tolerance to the procedure by means of a special analogue numerical scale checked after patient's awakening from anesthesia at the end of the intervention.
* occurrence of any complications or adverse event during the procedure (desaturation episodes, hemodynamic changes, oral-pharynx and larynx traumatism)

The primary endpoint is the comparison of success rate for the tracheal intubation in patients with anticipated difficult airways, demonstrating the non inferiority of videostylet efficacy compare to the most consolidated technique based on videolaryngoscope.

The Null Hypothesis will be the following: The rate of Awake tracheal intubation failure with the VS video stylet is > 10% compared to video-laryngoscope.

Considering an unsuccessful intubation rate with the two devices at 10%, a sample of 34 patients (17 per group) is necessary to demonstrate with a power of 90% and alpha error of 0.05 that the rate of intubation failure using the videosylet (study method) does not exceed 10% of the rate of failed intubations through the use of the video laryngoscope (reference method).

Statistical analysis:

Normally distributed data will be expressed as mean ± standard deviation and 95% confidence interval, while data with non-normal distribution will be expressed as median and interquartile range.

The differences between means will be studied by parametric tests (e.g. Student's t) if the data are normally distributed and by nonparametric tests (e.g. Wilcoxon) if the distribution is not normal. The Kolmogorov-Smirnov test will be used to evaluate the normality of continuous variables.

The characteristics of the patients in the two groups will be compared using the Fisher test or the Chi-square test for the nominal variables and the Student t test or the Mann - Whitney U test for the continuous variables.

For each test p < 0.05 will be considered significant. For the primary endpoint: The difference in awake tracheal intubation success rate in the two groups will be assessed using Fisher's exact test. The non-inferiority of the use of the videostylet (VS) compared to the standard method (videolaryngoscope with D-Blade blade) will be confirmed if the difference, for 95% confidence interval, is less than the margin of non- inferiority established "a priori" as 10% after analysis of the literature (Alhomary et al. Anaesthesia 2018; 73: 1151-61)9 and according to clinical judgment.

For the secondary endpoints of the study a purely analytical-descriptive evaluation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Schedule for elective surgery
* Detection of one or more of the following anthropometric criteria predictive of difficult intubation at the preoperative visit:

  1. Limitation of Cervical spine movements (traumatic or surgical arthrodesis)
  2. Mallampati score = 4
  3. Thyromental distance < 6 cm
  4. Interincisor distance < 3 cm
  5. Suspected difficult ventilation via face mask
  6. Previous history of difficult or failed intubation

Exclusion Criteria:

* age <18 years
* refusal of the patient
* urgent-emergency surgery
* patient's respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
the success rate of the rigid fiberoptic stylet to perform tracheal intubation in patients with anticipated difficult airways | up to a maximum of 3 attempts and up to 3 minutes from device insertion for each attempt (max 9 minutes)
  The primary endopoint is the comparison of success rate for the tracheal intubation in patients with anticipated difficult airways, demonstrating the non inferiority of videostylet efficacy compare to the most consolidated technique based on videolaryngoscope.
  success rate of the procedure defined as correct positioning of the tracheal tube in the trachea confirmed both endoscopically and through the capnographic curve EtCO2

SECONDARY OUTCOMES:
Numbers of intubation attempts | up to a maximum of 3 attempts and up to 3 minutes from device insertion for each attempt (max 9 minutes)
  number of attempt to intubation. intubation will be considered complete when the ETT (endotracheal tube) will be positioned correctly into the trachea
average time of intubation procedure expressed in seconds | up to 15 minutes
  Time in minutes measured from device insertion into the patient's mouth until theETT will be positioned into the trachea
Development of any complications | up to 12 hours measured from the insertion of the device
  occurrence of any complications or adverse event during the procedure (desaturation episodes, hemodynamic changes, oral-pharynx and larynx traumatism)
The degree of patient's tolerability of the procedure (with a special Analogue Numerical Scale) | up to 12 hours from the beginning of the procedure (from starting of awake intubation to complete recovering from general anaesthesia)
  assessment of the patient's tolerance to the procedure by means of the Visual Numerical Scale checked after patient's awakening from anesthesia at the end of the intervention. The Numerical Analogue Scales is a measurement instrument for tolerance-intensity. it consists of a numerical line from 1 to 5 with the endpoints defining extreme limits that are 5="not possible to tolerate at all" and 1="easily tolerable". the patient is asked to mark his tolerance-level on the line between the two endpoints
The degree of subjective difficulty experienced by the operator | up to 15 minutes (from device insertion into the patient's mouth until the ETT will be positioned into the trachea)
  operator's assessment of the subjective difficulty / handling of the device by means of a special analogue numerical scale from 1 to 5, where 1=no subjective difficulty and 5=maximal subjective difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, PhD, MD, Study Director — Università Politecnica delle Marche
Locations (1):
- AOU Ospedali Riuniti Ancona - Università Politecnica delle Marche, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No